CLINICAL TRIAL: NCT03502226
Title: Evaluation of an Inpatient Sexual Risk Behavior Assessment Program
Acronym: iRAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Oh-Zopfi Pilot Award 2016-2017
Record Dates: First submitted 2018-04-04; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-03

CONDITIONS: Adolescent Behavior; Sexual Behavior
MeSH Terms: conditions — Adolescent Behavior; Sexual Behavior

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Received tailored feedback regarding sexual health risks
  Interventions: Behavioral: Tailored feedback
- Control group (No Intervention): Did not receive tailored feedback.

INTERVENTIONS:
Behavioral: Tailored feedback — Electronic feedback based on participants "stage of change" which provided risk reduction behavior regarding their sexual health including use of condoms, contraceptions, and STI testing.
  Arms: Intervention group

SUMMARY:
This is an exploratory pilot study to evaluate the feasibility and potential effects of an innovative, individualized electronic inpatient sexual health intervention (iRAP) for adolescent females. The central hypothesis is that the electronic intervention, a sexual health questionnaire with tailored feedback based on the Trans Theoretical Model (TTM) of behavior change, will significantly increase adolescent females' requests for sexually transmitted infection (STI) screening and sexual health management during their hospital admission.

DETAILED DESCRIPTION:
Sexually transmitted infections (STIs) are disproportionately common among 15-24 year-old females, and can have detrimental effects including pelvic inflammatory disease and infertility. Most STI's are asymptomatic, especially for females, making screening programs essential. Current guidelines recommend HIV screening for all adolescents, and yearly chlamydia and gonorrhea screening for sexually active females under 25 years-old. Yet only one-third of primary care physicians report screening asymptomatic adolescents. Most adolescents report no sexual health discussion during preventative healthcare visits. Furthermore the majority do not regularly attend preventative healthcare visits. Therefore, urgent healthcare visits, often in emergency departments (ED) and inpatient settings, provide an important point of contact.

Given adolescents infrequently obtain outpatient sexual health services, the inpatient stay may serve as a critical intervention point. Other studies have found success with STI screening programs in the ED; none to our knowledge examined the efficacy of an inpatient sexual health screening protocol. Previous pilot data demonstrated, however, significant interest in sexual health information and desire for STI testing among adolescents admitted to a children's hospital.

Investigators conducted an exploratory study to evaluate the feasibility and potential effects of an innovative, individualized electronic inpatient sexual health intervention (iRAP) for adolescent females. The central hypothesis is that the electronic intervention, based on the Trans Theoretical Model (TTM) of behavior change, will significantly increase adolescent females' requests for STI screening and sexual health management.

Investigators enrolled 70 14-18 year-old, medically stable female inpatients admitted to the hospitalist service at Hasbro Children's Hospital for a randomized control trial during a one-year period. Participants were randomized to receive an electronic sexual risk assessment with or without real-time tailored feedback. Feedback was based on the TTM, utilizing readiness for change to determine appropriate messaging. Participants were then able to electronically request sexual health management options, including STI testing, discussion with their inpatient or outpatient physician, or technology-hosted information on contraception. Investigators conducted a chart review of enrolled adolescents to determine if sexual health topics were addressed.

The investigators are examining participation rates, length of time to perform all study elements, and proportion of teens that obtain requested service. Additionally, the investigators are comparing participants' perceived reproductive health risk and uptake of offered services between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Hospitalist service, English speaking, parent available for consent, medically/psychologically stable.

Exclusion Criteria:

* Wards of the state, no parent/guardian for consent, non-English speaking

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2017-10-29 (Actual); Study Completion 2017-10-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with requests for sexual health services, as assessed by sexual health options questionnaire | Immediate
  All participants were able to request sexual health services while admitted to the hospital (options included: STI testing, speak with their MD, or watching contraception video). The services were offered using an electronic REDCap questionnaire, with prompt of "Would you like to request X during your hospital stay?" and response options of yes/no. The outcome will be assessed for each sexual health option (number of participants requesting STI testing, discussion with MD, or contraception video viewing) individually, as well as a variable created to show "any uptake" ie. request made for any one or more services.